CLINICAL TRIAL: NCT00019955
Title: A Phase II Study to Evaluate Radiofrequency Ablation of Renal Cancer
Brief Title: Radiofrequency Interstitial Tissue Ablation in Treating Patients With Localized Renal Cell Carcinoma (Kidney Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067334; NCI-99-C-0170; NCT00001834 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2005-09

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Laparoscopy; Radiofrequency Ablation

INTERVENTIONS:
Procedure: laparoscopic surgery
Procedure: radiofrequency ablation
Procedure: thermal ablation therapy

SUMMARY:
RATIONALE: Radiofrequency interstitial tissue ablation may kill tumor cells by heating tumors to several degrees above body temperature.

PURPOSE: This phase II trial is studying radiofrequency interstitial tissue ablation to see how well it works in treating patients with localized renal cell carcinoma (kidney cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of radiofrequency interstitial tissue ablation in terms of tumor destruction or slowed tumor growth rate in patients with localized renal cell carcinoma.

Secondary

* Assess the toxicity of this treatment regimen in these patients.

OUTLINE: Patients undergo percutaneous radiofrequency interstitial tumor ablation (RFA). Patients are offered laparoscopy-assisted percutaneous RFA in the operating room if their tumors are not safely accessible. Intra-operative ultrasound is used to confirm probe placement and to monitor treatment delivery. If the target temperature or impedance are not reached, treatment is repeated no more than twice. No more than 5 tumors are treated per kidney.

All patients are followed at 2 to 3 months, 6 months, and then at 1 year.

Patients with tumors greater than 2 cm in diameter are followed every 6 months for up to 5 years. Patients whose tumors become greater than 3 cm are recommended for surgery and removed from study if surgery is performed.

PROJECTED ACCRUAL: A total of 63 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Localized renal cell carcinoma, meeting both of the following criteria:

  * Enlarging renal tumors on imaging studies over a minimum of 12 months
  * Tumor size between 0.5-4.0 cm in diameter at time of treatment

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine less than 2.0 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Other:

* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specifed

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03

PRIMARY OUTCOMES:
Response

CONTACTS AND LOCATIONS:
Overall Officials: McClellan M. Walther, MD, Study Chair — NCI - Urologic Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hwang JJ, Walther MM. Update on minimally invasive approaches to kidney tumors. Curr Urol Rep. 2004 Feb;5(1):13-8. doi: 10.1007/s11934-004-0005-y. PMID 14733831
- [Background] Pautler SE, Walther MM. Transperitoneal laparoscopic radical nephrectomy for bulky renal tumors. Can J Urol. 2002 Oct;9(5):1653-9; discussion 1660. PMID 12431330
- [Background] Pavlovich CP, Walther MM, Eyler RA, Hewitt SM, Zbar B, Linehan WM, Merino MJ. Renal tumors in the Birt-Hogg-Dube syndrome. Am J Surg Pathol. 2002 Dec;26(12):1542-52. doi: 10.1097/00000478-200212000-00002. PMID 12459621
- [Background] Wood BJ, Ramkaransingh JR, Fojo T, Walther MM, Libutti SK. Percutaneous tumor ablation with radiofrequency. Cancer. 2002 Jan 15;94(2):443-51. doi: 10.1002/cncr.10234. PMID 11900230
- [Background] Friedman M, Mikityansky I, Kam A, Libutti SK, Walther MM, Neeman Z, Locklin JK, Wood BJ. Radiofrequency ablation of cancer. Cardiovasc Intervent Radiol. 2004 Sep-Oct;27(5):427-34. doi: 10.1007/s00270-004-0062-0. Epub 2004 Jun 3. PMID 15383844
- [Background] Pautler SE, Pavlovich CP, Mikityansky I, Drachenberg DE, Choyke PL, Linehan WM, Wood BJ, Walther MM. Retroperitoneoscopic-guided radiofrequency ablation of renal tumors. Can J Urol. 2001 Aug;8(4):1330-3. PMID 11564277
- [Background] Kam AW, Littrup PJ, Walther MM, Hvizda J, Wood BJ. Thermal protection during percutaneous thermal ablation of renal cell carcinoma. J Vasc Interv Radiol. 2004 Jul;15(7):753-8. doi: 10.1097/01.rvi.0000133535.16753.58. PMID 15231890
- [Background] Pacak K, Fojo T, Goldstein DS, Eisenhofer G, Walther MM, Linehan WM, Bachenheimer L, Abraham J, Wood BJ. Radiofrequency ablation: a novel approach for treatment of metastatic pheochromocytoma. J Natl Cancer Inst. 2001 Apr 18;93(8):648-9. doi: 10.1093/jnci/93.8.648. No abstract available. PMID 11309443
- [Result] Hwang JJ, Walther MM, Pautler SE, Coleman JA, Hvizda J, Peterson J, Linehan WM, Wood BJ. Radio frequency ablation of small renal tumors:: intermediate results. J Urol. 2004 May;171(5):1814-8. doi: 10.1097/01.ju.0000119905.72574.de. PMID 15076283
- [Result] Pavlovich CP, Walther M, Choyke PL, Pautler SE, Chang R, Linehan WM, Wood BJ. Percutaneous radio frequency ablation of small renal tumors: initial results. J Urol. 2002 Jan;167(1):10-5. PMID 11743264
- [Result] Walther MC, Shawker TH, Libutti SK, Lubensky I, Choyke PL, Venzon D, Linehan WM. A phase 2 study of radio frequency interstitial tissue ablation of localized renal tumors. J Urol. 2000 May;163(5):1424-7. PMID 10751849